CLINICAL TRIAL: NCT01267695
Title: Perioperative Imatinib Mesylate in Treating Patients With Locally Advanced Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Ziyu Li, vice director of Department of Gastrointestinal Surgery，Peking University Cancer Hospital and Institute, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WJP-320.6700.09010
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: Gastrointestinal Stromal Tumor; Imatinib mesylate; Perioperative therapy
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: imatinib mesylate — Patients receive oral imatinib mesylate once daily for 6 months in the absence of disease progression or unacceptable toxicity. Patients with disease progression or unacceptable toxicity are considered for immediate surgical resection. Within 2-6 weeks after completion of imatinib mesylate, patients with responding or stable disease undergo surgical resection. Two to four weeks after surgery, patients receive oral imatinib mesylate once daily for one and a half years.
  Other Names: Gleevec; STI-571; NSC #716051
Procedure: conventional surgery — All the patients should receive elective surgery with R0 resection.

SUMMARY:
Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Perioperative imatinib mesylate may shrink the tumor and may reduce the chance of relapse after surgery. This phase II trial is studying the effectiveness of perioperative imatinib mesylate in treating patients with locally advanced gastrointestinal stromal tumor.

DETAILED DESCRIPTION:
Open-label trial in patients with locally advanced GISTs admitted to Department of Surgery, Beijing Cancer Hospital and Institute between April 2010 and May 2013 was carried out prospectively. Patients were planned to be treated with imatinib for duration of 6 months followed by surgical resection. Postoperative imatinib was planned to be administrated for 1.5 years. The primary end point was recurrent free survival (RFS) at 2 years; the secondary end points included objective response rate (ORR), surgical outcomes and drug safety.

ELIGIBILITY:
Criteria:

* DISEASE CHARACTERISTICS:

  * Histologically confirmed gastrointestinal stromal tumor

    * Locally advanced disease: tumour size >5 cm and mitotic count >5/HPF; tumour size >10 cm; mitotic count >10/HPF
    * Potentially resectable disease: Multivisceral resection may be necessary to get sufficient margins
  * Documented c-kit (CD117) expression by immunohistochemical analysis of either initial core specimen or, if recurrent disease, from original tumor block
  * At least 1 site of measurable disease
  * No known brain metastases
* PATIENT CHARACTERISTICS:

Age:18 and over Performance status:ECOG 0-3 Life expectancy:Not specified

* Platelet count > 100,000/mm3
* Absolute neutrophil count > 1,500/mm3 Hepatic
* AST and ALT < 2.5 times upper limits of normal (ULN) (5 times ULN if hepatic metastases are present)
* Bilirubin < 1.5 times ULN
* No chronic active hepatitis
* No cirrhosis
* No other chronic liver disease Renal
* Creatinine < 1.5 times ULN
* No chronic renal disease Cardiovascular
* No New York Heart Association class III-IV cardiac disease
* No congestive heart failure
* No myocardial infarction within the past 6 months Immunology
* No active uncontrolled infection
* No known HIV positivity Other
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* Must be medically fit to undergo surgery
* No other primary malignancy within the past 5 years except basal cell skin cancer, carcinoma in situ of the cervix, or a primary malignancy that is not currently clinically significant and does not require active intervention
* No gastrointestinal obstruction or major bleeding episode requiring immediate surgical intervention
* No uncontrolled diabetes
* No other severe or uncontrolled medical disease
* No significant history of noncompliance to medical regimens

PRIOR CONCURRENT THERAPY:

* No concurrent anticancer biologic agents
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) unless disease is rapidly progressing
* No concurrent anticancer chemotherapy
* At least 28 days since prior radiotherapy
* More than 2 weeks since prior major surgery except tumor biopsy Other
* At least 28 days since prior investigational drugs
* At least 28 days since prior imatinib mesylate
* No concurrent therapeutic doses of warfarin
* Concurrent low-molecular weight heparin or mini-dose warfarin (1 mg per day) prophylaxis is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Rate of disease recurrence at 2 years | 4 years

SECONDARY OUTCOMES:
Rates of objective response (complete, partial, and stable) | 2 years
Determine the safety and tolerability of this drug in these patients. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University School of Oncology, Beijing, China

REFERENCES:
- [Background] Eisenberg BL, Harris J, Blanke CD, Demetri GD, Heinrich MC, Watson JC, Hoffman JP, Okuno S, Kane JM, von Mehren M. Phase II trial of neoadjuvant/adjuvant imatinib mesylate (IM) for advanced primary and metastatic/recurrent operable gastrointestinal stromal tumor (GIST): early results of RTOG 0132/ACRIN 6665. J Surg Oncol. 2009 Jan 1;99(1):42-7. doi: 10.1002/jso.21160. PMID 18942073
- [Background] Seshadri RA, Rajendranath R. Neoadjuvant imatinib in locally advanced gastrointestinal stromal tumors. J Cancer Res Ther. 2009 Oct-Dec;5(4):267-71. doi: 10.4103/0973-1482.59905. PMID 20160360
- [Background] Saied GM, Kensarah AM. Six months neoadjuvant imatinib improves resectability potential of gastric stromal tumors in Egyptian patients. Int J Surg. 2010;8(2):105-8. doi: 10.1016/j.ijsu.2009.09.016. Epub 2009 Nov 24. PMID 19944196
- [Background] Machlenkin S, Pinsk I, Tulchinsky H, Ziv Y, Sayfan J, Duek D, Rabau M, Walfisch S. The effect of neoadjuvant Imatinib therapy on outcome and survival after rectal gastrointestinal stromal tumour. Colorectal Dis. 2011 Oct;13(10):1110-5. doi: 10.1111/j.1463-1318.2010.02442.x. PMID 21040362
- See also: Related Info — http://www.uptodate.com/patients/content/topic.do?topicKey=~1ahlhQH65OZROGa